CLINICAL TRIAL: NCT00273351
Title: Assessment of Pre-symptomatic and Symptomatic Patients With Parkinson Disease to Identify and Characterize Genetic and Phenotypic Biomarkers for Disease Onset and Progression.
Brief Title: Imaging and Genetic Biomarkers of Parkinson Disease (PD) Onset and Progression in High-risk Families
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Molecular NeuroImaging (Other)
Responsible Party: Principal Investigator, Kenneth Marek, MD, Principal Investigator, Institute for Neurodegenerative Disorders
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PROSPECT
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Parkinson Disease; Parkinsonian Syndrome
Keywords: Parkinson; family history; diagnosis
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [123I]B-CIT (Experimental): [123I]B-CIT and SPECT imaging
  Interventions: Drug: [123I]B-CIT

INTERVENTIONS:
Drug: [123I]B-CIT — Subjects will receive up to 6 mCi of [123I] B-CIT injected intravenously

SUMMARY:
Parkinson's disease (PD) is a progressive neurodegenerative disorder characterized by rigidity, bradykinesia, postural instability, and tremor. Clinical decline reflects ongoing degeneration of dopamine-containing neurons. A critical unmet need for clinical research is to improve early detection of these diseases by developing tools to assist with earlier diagnosis. Biomarkers are broadly defined as characteristics that are objectively measured and evaluated as indicators of normal biological processes, pathogenic processes, or pharmacologic responses to a therapeutic intervention (Biomarkers Defintions Working Group 2001). Development of reliable biomarkers for PD would dramatically accelerate research on PD etiology, pathophysiology, disease progression and therapeutics. Specific biomarkers may be useful at the onset of neurodegeneration, the onset of disease, and/or to mark disease progression. The biomarkers in this study include brain imaging with a radioactively labelled drug (Beta-CIT), computerized testing of memory, attention, motor speed, judgment and handwriting, and assessments of speech and smell. Subjects may also be asked to provide a blood sample for genetic and biochemical testing.

DETAILED DESCRIPTION:
Individuals who agree to participate in this trial will have a complete screening exam by a neurologist at the Institute for Neurodegenerative Disorders (IND) in New Haven, CT. The exam may include blood tests, urine tests and an electrocardiogram (ECG -tracing of the electrical activity of the heart) to determine eligibility for the trial.

Research subjects will participate in a variety of biomarker assessments including brain imaging, which will take place over a period of two days.

On the first day subjects report to IND after a brief exam subjects will receive a standard dose of Lugol's solution (potassium iodide) by mouth to decrease uptake of the radioactive drug into the thyroid gland. Subjects will be given a standard dose of potassium perchlorate if allergic to iodine.

Next subjects will receive the intravenous (IV - into a vein) injection of the Beta-CIT, a radioactive material that localizes in the brain.

On the second day, about 24 hours after the injection, subjects will return to IND for a SPECT scan. The SPECT camera takes a "picture" of the radiation emitted by the Beta-CIT. This procedure will take approximately 30 minutes.

Subjects will be contacted by phone one week following the injection to monitor adverse (bad or harmful) events possibly related to the imaging procedure.

This two-day imaging procedure, comprehensive neurological testing, and blood collection for genetics and biochemical testing may be repeated every 12 to 18 months during the next five years.

ELIGIBILITY:
Inclusion Criteria:

* Age >21
* Previous participation in the Progeni or Core PD clinical study
* A diagnosis of parkinsonism or a family history of parkinsonism
* Normal screening laboratory studies including:
* complete blood count
* chemistries
* urinalysis

Exclusion Criteria:

* Pregnancy
* Psychiatric disease other than history of depression
* Significant medical disease including abnormalities on screening biochemical or hematological labs or abnormal ECG.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2006-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Dopamine transporter density | 4.5 years
  The dopamine transporter density in individuals at risk for Parkinsonism due to family history compared to healthy controls.

SECONDARY OUTCOMES:
Correlation of the imaging outcome with both clinical outcomes (olfaction, reaction time, handwriting, etc) and biochemical measures | 4.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L. Marek, MD, Principal Investigator — President and Senior Scientist
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States

REFERENCES:
- [Background] Autere JM, Hiltunen MJ, Mannermaa AJ, Jakala PA, Hartikainen PH, Majamaa K, Alafuzoff I, Soininen HS. Molecular genetic analysis of the alpha-synuclein and the parkin gene in Parkinson's disease in Finland. Eur J Neurol. 2002 Sep;9(5):479-83. doi: 10.1046/j.1468-1331.2002.00458.x. PMID 12220378
- [Background] Foroud T, Uniacke SK, Liu L, Pankratz N, Rudolph A, Halter C, Shults C, Marder K, Conneally PM, Nichols WC; Parkinson Study Group. Heterozygosity for a mutation in the parkin gene leads to later onset Parkinson disease. Neurology. 2003 Mar 11;60(5):796-801. doi: 10.1212/01.wnl.0000049470.00180.07. PMID 12629236
- [Background] Golbe LI, Di Iorio G, Sanges G, Lazzarini AM, La Sala S, Bonavita V, Duvoisin RC. Clinical genetic analysis of Parkinson's disease in the Contursi kindred. Ann Neurol. 1996 Nov;40(5):767-75. doi: 10.1002/ana.410400513. PMID 8957018
- [Background] Kitada T, Asakawa S, Hattori N, Matsumine H, Yamamura Y, Minoshima S, Yokochi M, Mizuno Y, Shimizu N. Mutations in the parkin gene cause autosomal recessive juvenile parkinsonism. Nature. 1998 Apr 9;392(6676):605-8. doi: 10.1038/33416. PMID 9560156
- [Background] Koller WC, Langston JW, Hubble JP, Irwin I, Zack M, Golbe L, Forno L, Ellenberg J, Kurland L, Ruttenber AJ, et al. Does a long preclinical period occur in Parkinson's disease? Neurology. 1991 May;41(5 Suppl 2):8-13. No abstract available. PMID 2041599
- [Background] Lincoln SJ, Maraganore DM, Lesnick TG, Bounds R, de Andrade M, Bower JH, Hardy JA, Farrer MJ. Parkin variants in North American Parkinson's disease: cases and controls. Mov Disord. 2003 Nov;18(11):1306-11. doi: 10.1002/mds.10601. PMID 14639672
- [Background] Marek, K., J. Seibyl, et al. (1999). "[123I] ß-CIT/SPECT: Assessment of determinants of variability in progression of Parkinson's disease." Neurology 52: A91-92.
- [Background] Marek, K., J. Seibyl, et al. (1996). "Dopamine transporter and receptor imaging in Parkinsonism. (Presented at the 4th International Congress of Movement Disorders, Vienna, Austria; June, 1996.)." Mov Dis 6.
- [Background] Polymeropoulos MH, Higgins JJ, Golbe LI, Johnson WG, Ide SE, Di Iorio G, Sanges G, Stenroos ES, Pho LT, Schaffer AA, Lazzarini AM, Nussbaum RL, Duvoisin RC. Mapping of a gene for Parkinson's disease to chromosome 4q21-q23. Science. 1996 Nov 15;274(5290):1197-9. doi: 10.1126/science.274.5290.1197. PMID 8895469
- [Background] Seibyl JP, Marek KL, Quinlan D, Sheff K, Zoghbi S, Zea-Ponce Y, Baldwin RM, Fussell B, Smith EO, Charney DS, van Dyck C, et al. Decreased single-photon emission computed tomographic [123I]beta-CIT striatal uptake correlates with symptom severity in Parkinson's disease. Ann Neurol. 1995 Oct;38(4):589-98. doi: 10.1002/ana.410380407. PMID 7574455
- [Background] Seibyl JP, Marek K, Sheff K, Baldwin RM, Zoghbi S, Zea-Ponce Y, Charney DS, van Dyck CH, Hoffer PB, Innis RB. Test/retest reproducibility of iodine-123-betaCIT SPECT brain measurement of dopamine transporters in Parkinson's patients. J Nucl Med. 1997 Sep;38(9):1453-9. PMID 9293807
- [Background] Seibyl, J. P., K. L. Marek, et al. (1994). "[123I] B-CIT SPECT imaging in idiopathic parkinson's disease: correlation of striatal binding abnormality with disease severity [abstract]." Mov Disord 9(Suppl 1): 89.
- [Background] Tanner, C. (1994). Epidemiologic clues to the cause of Parkinson's disease. Movement Disorders 3. S. Fahn and C. Marsden. Oxford, Butterworth-Heinemann: 124-146.
- [Background] van Dyck CH, Seibyl JP, Malison RT, Laruelle M, Wallace E, Zoghbi SS, Zea-Ponce Y, Baldwin RM, Charney DS, Hoffer PB. Age-related decline in striatal dopamine transporter binding with iodine-123-beta-CITSPECT. J Nucl Med. 1995 Jul;36(7):1175-81. PMID 7790941
- [Background] Vingerhoets FJ, Snow BJ, Lee CS, Schulzer M, Mak E, Calne DB. Longitudinal fluorodopa positron emission tomographic studies of the evolution of idiopathic parkinsonism. Ann Neurol. 1994 Nov;36(5):759-64. doi: 10.1002/ana.410360512. PMID 7979222
- [Background] West AB, Maraganore D, Crook J, Lesnick T, Lockhart PJ, Wilkes KM, Kapatos G, Hardy JA, Farrer MJ. Functional association of the parkin gene promoter with idiopathic Parkinson's disease. Hum Mol Genet. 2002 Oct 15;11(22):2787-92. doi: 10.1093/hmg/11.22.2787. PMID 12374768